CLINICAL TRIAL: NCT04585841
Title: The Effect of Medical Cannabidiol on Lean Body Mass in Patients Receiving Oxaliplatin or Paclitaxel Based Chemotherapy
Brief Title: The Effect of Cannabidiol on Lean Body Mass in Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-846
Record Dates: First submitted 2020-09-10; First posted 2020-10-14 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Lean Body Mass; Cannabis; Cancer; Nausea; Cachexia; Emesis; Appetitive Behavior
Keywords: Cannabidiol; Cancer cachexia; Nausea; Emesis; Lean Body Mass; Oxaliplatin; Paclitaxel; Appetite; Adult; Quality of life; Taste alteration
MeSH Terms: conditions — Marijuana Abuse; Neoplasms; Nausea; Cachexia; Vomiting; Appetitive Behavior; Dysgeusia | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Cancer patients entering a phase 2 trial on cannabis for prevention on chemotherapy-induced peripheral neuropathy are asked to enter this study monitoring cannabidiols effect on lean body mass during chemotherapy. 40 participants are expected to enter intervention group, 20 participants in control group.
Masking Description: Control group will enter this study if not wanting to participate in cannabidiol study. Due to this masking is not possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cancer patients receiving cannabidiol
  Interventions: Drug: Cannabidiol
- Control group (No Intervention): Cancer patients not receiving cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Patients will receive cannabidiol in the period of time they receive chemotherapy.
  Other Names: No intervention
  Arms: Intervention group

SUMMARY:
An intervention study on the effect of cannabidiol on lean body mass in cancer patients receiving chemotherapy, at the department of Clinical Oncology at Zealand University Hospital, Roskilde, Denmark. Fat free mass will be measured by bioimpedance spectroscopy. As secondary outcomes protein and energy intake, nausea, taste alterations and life quality will be assessed by oral interviews and questionnaires.

DETAILED DESCRIPTION:
One of the side effects of chemotherapy is loss of lean body mass. With a non-blinded two armed intervention design this study will examine the effect of cannabidiol on fat free mass in cancer patients. The study will include patients who are diagnosed with cancer and scheduled to undergo at least 4 courses of paclitaxel or oxaliplatin based chemotherapy.

The hypothesis is that patients receiving cannabidiol (300mg/day) will have no change in lean body mass at the end of the study. In extension to this, we hypothesize that cannabidiol will increase the energy and protein intake because of increased appetite and decreased nausea and emesis.

Recruitment and data collection will take place at the department of Clinical Oncology at Zealand University Hospital, Roskilde.

Each patient will be included for four courses of paclitaxel or oxaliplatin based chemotherapy. The length between each chemotherapy course is three weeks.

Lean body mass will be measured by impedance spectroscopy before every chemotherapy treatment.

For two and a half months, patients will answer a weekly questionnaire about nausea, appetite and quality of life in general. The questionnaire is developed for this study.

In addition to the questionnaire, the patients will be interviewed about their daily dietary intake to quantify their energy and protein intake, calculated as percentage of estimated need.

Another side effect of chemotherapy is alterations in taste. In this study, we will examine the patient's taste in sweet and salty. At the day of chemotherapy, the patients will have a taste test. In the taste test the patients must tell which of the basic flavors they presume they are consuming, as well as how strong the taste is , on a scale from 1 to 10.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer
* Fulfill criteria for starting chemotherapy
* Must be able to stand upright
* Have the possibility of contact by telephone
* No previous treatment with taxanes or platinums
* Scheduled to undergo lest 4 courses of paclitaxel or 4 courses of oxaliplatin based chemotherapy
* If female and fertile, must have been menopausal for 1 year or negative pregnancy test at inclusion and use approved contraceptive measures

Exclusion Criteria:

* Pregnant
* Breastfeeding
* Unable to complete patient reported outcomes (PRO)-measurements
* Previously received taxanes or platinum-based chemotherapy
* Use of cannabinoids. If in use, treatment must be stopped 4 days prior to inclusion
* If using any anti epileptic or antidepressant medicine. Treatment must be stable (no changes in dosing in last 30 days) prior to inclusion. However, any treatment with Clobazam is not allowed due to major interaction with cannabidiol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with change in lean body mass from baseline. | 10 weeks
  Changes in lean body mass measured at baseline and before each chemotherapy treatment (scheduled for every three weeks) measured in kg by bioimpedance. Changes are assessed as change in percentage of total lean body mass weight.

SECONDARY OUTCOMES:
Change in food intake | 10 weeks
  Change in food intake from baseline measured in kilojoule (kJ). Changes in intake of protein- and energy assessed by weekly nutritional recall interviews of weekly intake.
  Change in food intake from baseline measured in kJ. Changes in intake of protein- and energy assessed by weekly nutritional recall interviews of weekly intake.
Change in energy intake . | 10 weeks
  Change in intake of energy assessed by weekly nutritional 24-hour recall interview.
  Assessment of energy requirement using Harris Benedict- formula estimated from height in cm, weight in kilo, age in years and physical activity level (PAL). Height and weight is derived from bioimpedance measurements in Outcome 1. Age is derived from conversation with the participant. PAL is assessed after conversation with the participant. Energy requirements will be reported as kilojoule (Kj).
  Correlation between relative fulfilment of energy requirement, and change therein. Energy requirement is estimated by Harris-Benedict formula, including among other assessment of physical activity level.
Change in protein intake | 10 weeks
  Change in protein intake from baseline measured in kJ Protein requirement is estimated from the Danish Health Authority´s recommendation for adult patients. Protein intake is assessed by 24-hour recall of nutrition intake.
Change in nausea | 10 weeks
  Changes in nausea from baseline is assessed by a categorical scale in a weekly questionnaire if the participant is experiencing nausea: daily, five or six times a week, three or four times a week, one or two times a week, not at all. "Not at all" being the lowest score, "Daily" being the highest.
  The Questionnaire is written in danish and is called Livskvalitet (Quality of life) and the scale is for the question "Symptomer" (symptoms). The questionnaire is developed for this study and language validation has been done with 12 patients from the same department as the study will take place
Change in emesis | 10 weeks
  Changes in emesis from baseline is assessed by a categorical scale in a weekly questionnaire if the participant is experiencing nausea: daily, five or six times a week, three or four times a week, one or two times a week, not at all. "Not at all" being the lowest score, "Daily" being the highest.
  The Questionnaire is written in danish and is called Livskvalitet (Quality of life) and the scale is for the question "Symptomer" (symptoms). The questionnaire is developed for this study and language validation has been done with 12 patients from the same department as the study will take place.
Difference in taste during chemotherapy. | 10 weeks
  Difference in taste from baseline is measured by a sensory test with flavour neutral mashed potato added sweet, sour or umami flavour in two strengths of flavour. Participants will answer which flavour they taste and how strong the flavour is on a scale from 1-10. Also the patients preference in the three flavours will be monitored.
Change in appetite | 10 weeks
  Changes in appetite from baseline is assessed by a categorical scale in a weekly questionnaire about the patient's subjective estimation on portion size: bigger, the same or smaller than usual compared to the weekly nutritional 24-hour recall interview. Bigger being the highest value, smaller than usual being the lowest value.
Change in Quality of life (QOL) | 10 weeks
  To estimate the patient' QOL from baseline by a weekly questionnaire about the patient's well being. It will be compared with the questions about appetite, taste, nausea and emesis. It will also be compared with the patient medical record.
  The Questionnaire is written in danish and is called Livskvalitet (Quality of life) and the scale is for the question "Symptomer" (symptoms). The questionnaire is developed for this study and language validation has been done with 12 patients from the same department as the study will take place

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, Study Chair — University of Copenhagen; Sebastian W Nielsen, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark